CLINICAL TRIAL: NCT02675387
Title: Efficacy of External Cold and a Vibrating Device in Reducing Discomfort of Dental Injections in Children - A Split Mouth Randomized Clinical Trial
Brief Title: Efficacy of External Cold and a Vibrating Device in Reducing Discomfort of Dental Injections in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riyadh Colleges of Dentistry and Pharmacy (Other)
Responsible Party: Principal Investigator, Dr Sharat Pani, Program Director - Pediatric Dentistry, Riyadh Colleges of Dentistry and Pharmacy
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: FPGRP/43535001/163
Record Dates: First submitted 2016-01-18; First posted 2016-02-05 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Traditional Group (Active Comparator): Children will be administered buccal infiltration anesthesia using a 21mm needle and 1.8ml of 2%Lidocaine
  Interventions: Drug: 2%Lidocaine
- Buzzy (Experimental): Children will be administered buccal infiltration anesthesia using a 21mm needle and 1.8ml of 2%Lidocaine after sensitizing the area with a vibrating device
  Interventions: Device: Buzzy; Drug: 2%Lidocaine

INTERVENTIONS:
Device: Buzzy — Two minute application of a hand held vibrating device (Buzzy, MMJ labs, Atlanta GA, USA) before the administration of anesthesia
  Other Names: Vibrating Device
  Arms: Buzzy
Drug: 2%Lidocaine — 1.8ml of 2%Lidocaine HCl to be administered via a 21mm needle (30 Guage)
  Other Names: Lignocaine

SUMMARY:
Children in their seventh year of life (age range of 6 to 7 years) will be included in the study. All children included in the study would have to classified according to the Wright behavior classification as potentially co-operative and rated as per the Frankl behavior rating scale as positive (++) Group A and negative (-) Group B . All children included must have had no prior experience of dental anesthesia and must have at least one tooth requiring restorative procedure on either side of the maxillary arch. Intervention Description

1. Regular Anesthesia All the subjects received local anesthesia injection in maxillary arch as is commonly practiced in dental clinics. Information obtained before assignment of intervention or standard care included age, gender, type of injection given alongside the vibration device will be recorded beforehand. During the delivery of anesthesia for all the groups, anticipated and actual pain will be recorded to show the impact of anxiety on the experience of participants. During the entire process, all participants will use standard needles with confirmed specification to control for any potential confounders
2. Buzzy® The use of the external cold and a vibrating Device will follow the manufacturer's recommendations to ensure that normal clinical scenario is created.

DETAILED DESCRIPTION:
Methodology Ethical Clearance:The study will be registered at the clinical trials registry of the United States National Institutes of Health (NIH), following which ethical approval will be obtained from the institutional review board of the Riyadh Colleges of Dentistry and Pharmacy Patient Recruitment The sample will comprise of 60 children reporting to the clinics of the Riyadh Colleges of Dentistry and Pharmacy determine to have treatment that involve the use of local anesthesia.

Sample Power Calculation Sample power calculation was done using the G Power sample size calculator (Universtat Kiel, Kiel, Germany) . Given the split mouth study design proposed a high effect size of 0.8 was assumed. The minimum number of individuals for an alpha of 0.05 and a power of 0,95 was 19 subjects per group. Given the risk of attrition of subjects in the study, the total sample size recruited will be 30 per group (n=60)

The Inclusion Criteria Children in their seventh year of life (age range of 6 to 7 years) will be included in the study. All children included in the study would have to classified according to the Wright behavior classification as potentially co-operative and rated as per the Frankl behavior rating scale as positive (++) Group A and negative (-) Group B . All children included must have had no prior experience of dental anesthesia and must have at least one tooth requiring restorative procedure on either side of the maxillary arch. The classification of each patient will be done separately by two experienced pediatric dentists (NG and SCP) and consensus on the classification will be obtained before including the patient in the study. Informed consent will be obtained from the parent of all patients who agree to participate in the study.

Exclusion Criteria Patients with a history of hospitalization or surgery, those with chronic illness will be excluded from the study. The study will also exclude patients diagnosed with neurobehavioral disorders such as autism, ADHD or learning disability. Patients with congenital syndromes or intellectual disability will also be excluded from the study.

Intervention Description

1. Regular Anesthesia All the subjects received local anesthesia injection in maxillary arch as is commonly practiced in dental clinics. Information obtained before assignment of intervention or standard care included age, gender, type of injection given alongside the vibration device will be recorded beforehand. During the delivery of anesthesia for all the groups, anticipated and actual pain will be recorded to show the impact of anxiety on the experience of participants. During the entire process, all participants will use standard needles with confirmed specification to control for any potential confounders
2. Buzzy® The use of the external cold and a vibrating Device will follow the manufacturer's recommendations to ensure that normal clinical scenario is created.

ELIGIBILITY:
Inclusion Criteria:

* No prior experience of dental anesthesia
* At least one upper tooth on either side requiring anesthesia before restoration

Exclusion Criteria:

* History of mental illness
* Extensive hospitalization for chronic illness
* Past history of surgery

Ages: 6 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-03 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Pain of injection ( Wong Baker Face Pain Scale) | 0 min - at the time of injection
  Pain felt on injection measured using the Wong Baker Face Pain Scale
Pain of injection ( Wong Baker Face Pain Scale) | 5 min after the injection
  Pain felt measured using the Wong Baker Face Pain Scale
Pain of injection ( Wong Baker Face Pain Scale) | 30 min after the injection
  Pain felt measured using the Wong Baker Face Pain Scale

SECONDARY OUTCOMES:
Behavior ( Frankl behavior rating scale) | 5min before procedure, 5 min after completion of procedure
  Behavior measured using the Frankl behavior rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Sharat C Pani, Principal Investigator — Riyadh Colleges of Dentistry and Pharmacy
Locations (1):
- Riyadh Colleges of Dentistry and Pharmacy, Riyadh, Al Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Baxter AL, Lawson ML. Methodological concerns comparing buzzy to transilluminator device. Indian J Clin Biochem. 2014 Jan;29(1):114-5. doi: 10.1007/s12291-013-0370-8. Epub 2013 Sep 3. No abstract available. PMID 24478562
- [Result] Shahidi Bonjar AH. Syringe micro vibrator (SMV) a new device being introduced in dentistry to alleviate pain and anxiety of intraoral injections, and a comparative study with a similar device. Ann Surg Innov Res. 2011 Jan 7;5(1):1. doi: 10.1186/1750-1164-5-1. PMID 21211061
- [Result] Canbulat N, Ayhan F, Inal S. Effectiveness of external cold and vibration for procedural pain relief during peripheral intravenous cannulation in pediatric patients. Pain Manag Nurs. 2015 Feb;16(1):33-9. doi: 10.1016/j.pmn.2014.03.003. Epub 2014 Jun 7. PMID 24912740
- [Result] Canbulat Sahiner N, Inal S, Sevim Akbay A. The effect of combined stimulation of external cold and vibration during immunization on pain and anxiety levels in children. J Perianesth Nurs. 2015 Jun;30(3):228-35. doi: 10.1016/j.jopan.2014.05.011. PMID 26003770
- [Result] Czarnecki ML, Turner HN, Collins PM, Doellman D, Wrona S, Reynolds J. Procedural pain management: a position statement with clinical practice recommendations. Pain Manag Nurs. 2011 Jun;12(2):95-111. doi: 10.1016/j.pmn.2011.02.003. Epub 2011 Apr 29. PMID 21620311
- [Result] Jalevik B, Klingberg G. Pain sensation and injection techniques in maxillary dento-alveolar surgery procedures in children--a comparison between conventional and computerized injection techniques (The Wand). Swed Dent J. 2014;38(2):67-75. PMID 25102717
- [Result] Kandiah P, Tahmassebi JF. Comparing the onset of maxillary infiltration local anaesthesia and pain experience using the conventional technique vs. the Wand in children. Br Dent J. 2012 Nov;213(9):E15. doi: 10.1038/sj.bdj.2012.988. PMID 23138830
- [Result] Kearl YL, Yanger S, Montero S, Morelos-Howard E, Claudius I. Does Combined Use of the J-tip(R) and Buzzy(R) Device Decrease the Pain of Venipuncture in a Pediatric Population? J Pediatr Nurs. 2015 Nov-Dec;30(6):829-33. doi: 10.1016/j.pedn.2015.06.007. Epub 2015 Jul 27. PMID 26228308
- [Result] Nanitsos E, Vartuli R, Forte A, Dennison PJ, Peck CC. The effect of vibration on pain during local anaesthesia injections. Aust Dent J. 2009 Jun;54(2):94-100. doi: 10.1111/j.1834-7819.2009.01100.x. PMID 19473149
- [Result] Roeber B, Wallace DP, Rothe V, Salama F, Allen KD. Evaluation of the effects of the VibraJect attachment on pain in children receiving local anesthesia. Pediatr Dent. 2011 Jan-Feb;33(1):46-50. PMID 21406147
- [Result] Whelan HM, Kunselman AR, Thomas NJ, Moore J, Tamburro RF. The impact of a locally applied vibrating device on outpatient venipuncture in children. Clin Pediatr (Phila). 2014 Oct;53(12):1189-95. doi: 10.1177/0009922814538494. Epub 2014 Jun 12. PMID 24924565
- [Result] Wiederhold MD, Gao K, Wiederhold BK. Clinical use of virtual reality distraction system to reduce anxiety and pain in dental procedures. Cyberpsychol Behav Soc Netw. 2014 Jun;17(6):359-65. doi: 10.1089/cyber.2014.0203. PMID 24892198
- [Derived] Alanazi KJ, Pani S, AlGhanim N. Efficacy of external cold and a vibrating device in reducing discomfort of dental injections in children: A split mouth randomised crossover study. Eur Arch Paediatr Dent. 2019 Apr;20(2):79-84. doi: 10.1007/s40368-018-0399-8. Epub 2018 Dec 5. PMID 30519955